CLINICAL TRIAL: NCT02285452
Title: Psychophysiological Efficacy of Thorax Wraps With Ginger or Mustard Flour in Comparison to Wraps With Warm Water in Healthy Subjects - a Randomized, Placebo-controlled, Three-armed Study With Cross-over Design
Brief Title: Psychophysiological Effects of Thorax Wraps With Ginger and Mustard Flour
Acronym: SWI_02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: SWI_02
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: physiologcal phenomena; .HRV Parameters; respiratory activity; thorax wraps

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Thorax wrap with ginger flour (Zingiberis Rhizoma plv.) (Active Comparator): Thorax wrap with ginger flour, duration max. 20 minutes
  Interventions: Drug: Zingiberis Rhizoma plv.
- Thorax wrap with mustard flour (Sinapis nigrea semen) (Active Comparator): Thorax wrap with mustard flour, duration max 20 minutes
  Interventions: Drug: Sinapis nigrea semen
- Thorax wrap with warm water (placebo) (Placebo Comparator): Thorax wrap with warm water (placebo), duration: 20 minutes
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zingiberis Rhizoma plv.
  Arms: Thorax wrap with ginger flour (Zingiberis Rhizoma plv.)
Drug: Sinapis nigrea semen
  Arms: Thorax wrap with mustard flour (Sinapis nigrea semen)
Drug: Placebo
  Arms: Thorax wrap with warm water (placebo)

SUMMARY:
In integrative medicine wraps are applied for different indications. In this study the effects of thorax with ginger and mustard flour are investigated under standardized conditions. Heart rate variability, well being, warmth distribution and respiratory activity of healthy subjects will be measured.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effects of different thorax wraps in healthy subjects. Subjects undergo three different interventions (wraps with ginger flour, mustard flour or warm water (placebo)) on three different days. Heart rate variability and respiratory activity is measured for ten minutes before, during (up to 20 minutes) and for ten minutes after each thorax wrap. To investigate the effects on heat development and regulation, photos are taken with a thermographic infrared camera at various moments in time. Participants are asked to fill in questionnaires referring to their subjective perceptions of warmth, bodily warmth distribution and wellbeing. The order of the thorax wrap interventions is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.

Exclusion Criteria:

Inflectional disease with body temperature > 38 °C. Skin damage on the thorax area Known intolerance or hypersensitivity to mustard or ginger products. Heart failure. Asthma bronchiale. Taking medication with influence on heart rate variability ( mainly tricyclic antidepressants and beta blocker).

Consumption of coffee or nicotine less than three hours before the intervention.

Pregnancy. Deficient knowledge of the German language.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
changes in temperature | max. 40 minutes
  Temperature (in °Celsius) of feet, lower legs, hands and face measured with a thermographic infrared camera (pre-post-comparison)
Respiratory activity (expiratory CO2 and NO-measurement) | max. 40 minutes
  Physiological parameters are measured for pre-post comparison.

SECONDARY OUTCOMES:
Basler Mood Questionnaire (BBS) | 40 minutes
  filled in by the participants nine times (before and after the thorax wrap and 10 minutes after the intervention)
Herdecker Wärmeempfindungs-Fragebogen (HeWef) | 40 minutes
  filled in by the participants nine times (before and after the thorax wrap and 10 minutes after the intervention)
Warmth perception and skin irritation (NRS) | 40 minutes
  Warmth perception and skin irritation during the intervention every minute (measured with a numeric rating scale).
heart rate variability -Parameter (HRV) | Physiological parameters are measured over a period of 40 minutes
  Standard Deviation of Normal to Normal (heart rate) (SDNN)
heart rate variability -Parameter (HRV) | Physiological parameters are measured over a period of 40 minutes
  Root Mean Square of the Successive Differences (RMSSD)
heart rate variability -Parameter (HRV) | Physiological parameters are measured over a period of 40 minutes
  ratio low frequency to high frequency (LF/HF)
heart rate variability -Parameter (HRV) | Physiological parameters are measured over a period of 40 minutes
  very low frequency (VLF)
heart rate variability -Parameter (HRV) | Physiological parameters are measured over a period of 40 minutes
  NN50 (the number of pairs of successive NNs that differ by more than 50 ms)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr., Principal Investigator — ARCIM-Institute
Locations (1):
- Filderklinik, Filderstadt, Baden-Wurttemberg, Germany